CLINICAL TRIAL: NCT01404832
Title: The Frequency of Eosinophilic Esophagitis in Patients With Heartburn That is Refractory to Proton Pump Inhibitors
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Inadequate recruitment
Sponsor: Dallas VA Medical Center (U.S. Federal Agency)
Collaborators: TAP Pharmaceutical Products Inc. (Industry)
Responsible Party: Principal Investigator, Stuart Spechler, PI, Dallas VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VAIRB06-093
Record Dates: First submitted 2011-07-27; First posted 2011-07-28 (Estimated); Results first posted 2013-02-27 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Gastroesophageal Reflux Disease; Eosinophilic Esophagitis
Keywords: Gastroesophageal reflux; Proton pump inhibitor; Eosinophilic esophagitis
MeSH Terms: conditions — Gastroesophageal Reflux; Eosinophilic Esophagitis | interventions — Coal Tar; Lansoprazole; BID protein, human; Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Treat with lansoprazole 30 mg BID for 2 weeks, endoscopic examination with esophageal biopsy for patients with persistent symptoms — Treat with lansoprazole 30 mg BID for 2 weeks, perform endoscopic examination with esophageal biopsy

SUMMARY:
Background: Up to 40% of patients who are treated with PPIs for symptoms that are thought to be due to GERD experience only incomplete relief of their symptoms. Those patients are deemed "PPI failures." Esophageal pH monitoring studies have shown that PPI failure rarely is due to persistent acid reflux. Recently, heartburn that is refractory to treatment with PPIs has been described in patients with eosinophilic esophagitis, a disorder of unknown etiology in which eosinophils infiltrate the squamous epithelium of the esophagus, where they cause symptoms and tissue injury. Presently, it is not clear how often eosinophilic esophagitis underlies PPI failure for patients with GERD symptoms.

Purpose: To estimate the frequency with which eosinophilic esophagitis is the cause of "PPI failure" in patients thought to have heartburn due to GERD.

Methods: Patients referred to the Division of Gastroenterology at the Dallas VA Medical Center for the evaluation of heartburn that is refractory to PPI therapy will be invited to participate in the study. Patients who provide informed consent will have a medical history taken. Women of child bearing potential will have a pregnancy test. The patients' current PPI therapy will be discontinued, and patients will be treated with lansoprazole 30 mg BID for one week. The patient will return to the clinic one week later. Patients who feel that their heartburn has not improved by more than 50% from baseline will have an endoscopic evaluation. During the endoscopic examination, biopsy specimens will be taken as follows: A. Two specimens from the proximal esophagus at 20 cm from the incisor teeth. B. Two specimens from the mid-esophagus at 28 cm from the incisor teeth. C. Two specimens from the distal esophagus, 3 cm above the squamo-columnar junction. D. Two specimens from the distal esophagus, 1 cm above the squamo-columnar junction. E. Two specimens from the second portion of the duodenum (to see if the eosinophilia is confined to the esophagus, or part of a more extensive eosinophilic gastroenteritis). A diagnosis of eosinophilic esophagitis will be made if there is at least one high-power field with >25 eosinophils, or two or more high-power fields with >15 eosinophils.

Potential Benefits: This study will provide an estimate on the frequency with which eosinophilic esophagitis is the cause of "PPI failure" in patients thought to have heartburn due to GERD. This has substantial potential importance for patient management.

ELIGIBILITY:
Inclusion Criteria:Male and female patients ages 18 years and older who are referred to the Division of Gastroenterology at the Dallas VA Medical Center for the evaluation of heartburn that is refractory to PPI therapy

Exclusion Criteria:

1. Patients unwilling or unable to provide informed consent.
2. Allergy to lansoprazole.
3. Patients taking warfarin.
4. Coagulopathy that precludes safe biopsy of the esophagus.
5. Comorbidity that precludes safe participation in the study.
6. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2007-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart J Spechler, MD, Principal Investigator — Dallas VA Medical Center
Locations (1):
- Dallas VA Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consecutive patients referred to a general GI clinic at our VA hospital for the evaluation of PPI-resistant heartburn were invited to participate.
Pre-assignment Details: 102 patients agreed to participate. For 10 patients the symptom described was not consistent with heartburn and another 27 described heartburn that was not refractory to therapy. 65 patient had PPI-resistant heartburn; 33 were taking PPI incorrectly; 11 taking insufficient dose of omeprazole.
Groups:
- Patients Whose PPI Was Changed to Lansoprazole: In 21 patients taking omeprazole ≥80 mg/day, the PPI was changed to lansoprazole 30 mg BID before breakfast and dinner.
Period: Overall Study
Arm/Group | Patients Whose PPI Was Changed to Lansoprazole
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients Whose PPI Was Changed to Lansoprazole
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Eosinophilic Esophagitis
Time Frame: 8 weeks
Measure: Number; unit: participants
Arm/Group | Patients Whose PPI Was Changed to Lansoprazole
Number analyzed (Participants) | 21
participants | 0

2. Secondary Outcome: Number of Patients Who Had Resolution of Heartburn With Lansoprazole
Description: Resolution of heartburn defined as >50% improvement in symptoms
Time Frame: After 8 weeks of treatment
Measure: Number; unit: participants
Arm/Group | Patients Whose PPI Was Changed to Lansoprazole
Number analyzed (Participants) | 21
participants | 9

ADVERSE EVENTS:
Arm/Group | Patients Whose PPI Was Changed to Lansoprazole
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No